CLINICAL TRIAL: NCT05803733
Title: The Effect of Blood Flow Restrictive Exercise on Grip Strength and Upper Extremity Functions in Elderly Individuals
Brief Title: Blood Flow Rextriction Training in Upper Extremity of Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Medipol University (Other); Bahçeşehir University (Other)
Responsible Party: Principal Investigator, gizem ergezen, Gizem Ergezen, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: E-10840098-772.02-7706
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Exercise Training; Blood Flow Restriction Training; Geriatrics
Keywords: Blood Flow Restriction Training; geriatrics; performance; muscle strength

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (BFR) with low load resistance training (Experimental): Participants will have the routine rehabilitation protocol and as an addition participants will use a cuff placed proximal to the arm during upper extremity strengthening exercises. The cuff to be used is 175mm wide and 920mm long. After the cuff is placed, it will be inflated to the determined arterial occlusion pressure. The pressure will be adjusted to 50% of the BP in the arm during rest and increased to 60%. Exercises will be performed with the cuff inflated, at approximately 20-30% of 1RM. The first set will be 30 repetitions or at the limit of fatigue (maximum of 4/10), then three sets of 15 repetitions. The cuff will not be deflated for the 30 second rest between sets. A rehabilitation session will be held under the supervision of a physiotherapist. Exercise will be performed for 6 weeks with 3 sessions each week, with 1-2 days break between sessions.
  Interventions: Other: Blood flow restriction (BFR) with low load resistance training; Other: Routine strength training
- Control Group (Active Comparator): Participants only will have the rehabilitation protocol including general physiotherapeutic approaches such as range of motion exercises and strength training which is a daily part of their nursing home services.
  Interventions: Other: Routine strength training

INTERVENTIONS:
Other: Blood flow restriction (BFR) with low load resistance training — Combination of low load resistance exercise in the upper limb.
  Arms: Blood flow restriction (BFR) with low load resistance training
Other: Routine strength training — range of motion exercises and strength training

SUMMARY:
Our study aims to decrease independence by increasing upper extremity strength and performance by applying blood flow restrictive training, which has entered the literature as a new method, to the upper extremity in the elderly. The application will only be applied to the upper extremity and will last for 6 weeks.

DETAILED DESCRIPTION:
People are living longer now than in the past. The experience of old age in modern societies has gained importance with the prolongation of life expectancy. Over the years, the elderly lead to a decrease in physiological capacity and an increase in the risk of various diseases, resulting in a decrease in the functional capacity of the individual. Many physiological changes occur in the organism with advancing age. Muscle strength is an important determinant of healthy aging. It is known that the decrease in muscle mass and strength impairs body function and can have significant consequences for the individual, as well as increase economic costs. Impairment in function initially results in difficulties performing common daily activities such as carrying household items; however, when body strength falls below a clinically relevant threshold, mobility restriction increases and may affect independence in activities of basic daily living. Loss of independence requires support from caregivers; often leads to social withdrawal and adverse effects on well-being and quality of life. Muscle strength, function and mobility are the biggest determinants of independence. Handgrip strength is used in clinical practice, rehabilitation, and public health research to determine musculoskeletal function and assess frailty and disability.

The aim of our study is to determine the effect of BFRT applied to the upper extremity for 6 weeks on general function, hand grip strength, upper extremity functional status, activities of daily living and functionality for elderly individuals between the ages of 65-75. Our hypothesis is that BFR will increase upper extremity function and related activities of daily living and mobility by increasing hand grip strength in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 65 and over who are classified as advanced age according to the World Health Organization
* Volunteer basis

Exclusion Criteria:

* History of acute trauma to the hand or wrist
* Scrapped upper extremity
* Patients with symptoms of shoulder or elbow pain and rheumatoid arthritis,
* Those who have participated in upper extremity weight training training in the last 6 months,
* Those taking sedatives
* Upper extremity venous thrombosis,
* Being at high risk for cardiovascular conditions that interfere with exercise, unexplained chest pain or heart disease, fainting or dizziness during physical activity/exercise

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Range of Motion- ROM (shoulder flexion) | Baseline
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer will be placed on the greater tubercle of the humerus, the fixed arm will be placed parallel to the patient's axillary line, and the movable arm will be placed parallel to the lateral midline of the humerus. The patient will be asked to move his arm above his head without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion- ROM (shoulder flexion) | 6 weeks
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer will be placed on the greater tubercle of the humerus, the fixed arm will be placed parallel to the patient's axillary line, and the movable arm will be placed parallel to the lateral midline of the humerus. The patient will be asked to move his arm above his head without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion- ROM (shoulder flexion) | 12 weeks
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer will be placed on the greater tubercle of the humerus, the fixed arm will be placed parallel to the patient's axillary line, and the movable arm will be placed parallel to the lateral midline of the humerus. The patient will be asked to move his arm above his head without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion - ROM (shoulder abduction) | Baseline
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer is placed on the acromion, the fixed arm is parallel to the sternum and the columna vertebralis, and the movable arm is placed parallel to the anterior midline of the humerus. The patient will be asked to move his arm by opening it from the side of the body without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion - ROM (shoulder abduction) | 6 weeks
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer is placed on the acromion, the fixed arm is parallel to the sternum and the columna vertebralis, and the movable arm is placed parallel to the anterior midline of the humerus. The patient will be asked to move his arm by opening it from the side of the body without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion - ROM (shoulder abduction) | 12 weeks
  The patient will be positioned in the supine position, with the arms next to the trunk and the elbow in extension. The pivot point of the goniometer is placed on the acromion, the fixed arm is parallel to the sternum and the columna vertebralis, and the movable arm is placed parallel to the anterior midline of the humerus. The patient will be asked to move his arm by opening it from the side of the body without breaking his elbow, and the final angle will be recorded in degrees.
Range of Motion - ROM (shoulder external rotation) | Baseline
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point of the goniometer will be placed in the olecranon, its fixed arm parallel to the ground at the edge of the measuring bed, and its movable arm parallel to the 3rd metacarpal. The patient will be asked to move the forearm in the direction of the thumb without lifting the elbow from the bed, and the last angle will be recorded in degrees.
Range of Motion - ROM (shoulder external rotation) | 6 weeks
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point of the goniometer will be placed in the olecranon, its fixed arm parallel to the ground at the edge of the measuring bed, and its movable arm parallel to the 3rd metacarpal. The patient will be asked to move the forearm in the direction of the thumb without lifting the elbow from the bed, and the last angle will be recorded in degrees.
Range of Motion - ROM (shoulder external rotation) | 12 weeks
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point of the goniometer will be placed in the olecranon, its fixed arm parallel to the ground at the edge of the measuring bed, and its movable arm parallel to the 3rd metacarpal. The patient will be asked to move the forearm in the direction of the thumb without lifting the elbow from the bed, and the last angle will be recorded in degrees.
Range of Motion - ROM (shoulder internal rotation) | Baseline
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point, fixed arm and movable arm of the goniometer are positioned as in the shoulder external rotation measurement. The patient will be asked to move his forearm towards the bed in the direction of his little finger without lifting his elbow from the bed, and the last angle will be recorded in degrees.
Range of Motion - ROM (shoulder internal rotation) | 6 weeks
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point, fixed arm and movable arm of the goniometer are positioned as in the shoulder external rotation measurement. The patient will be asked to move his forearm towards the bed in the direction of his little finger without lifting his elbow from the bed, and the last angle will be recorded in degrees.
Range of Motion - ROM (shoulder internal rotation) | 12 weeks
  The patient will be positioned in the supine position with the shoulder 90° abduction and the elbow 90° flexion. The pivot point, fixed arm and movable arm of the goniometer are positioned as in the shoulder external rotation measurement. The patient will be asked to move his forearm towards the bed in the direction of his little finger without lifting his elbow from the bed, and the last angle will be recorded in degrees.
Grip strength | Baseline
  grip strength It will be evaluated with the JAMAR™ isometric dynamometer (National Institute for Health Research, Southampton), a device recommended by the American Association of Hand Therapists (ASTH). The participant is seated in a chair without an armrest, feet flat on the floor, the shoulder is adducted with neutral rotation, the elbow is positioned at 90° flexion and the forearm is neutral. The JAMAR™ handle is worn in the second position, which allows for balanced activation of the intrinsic and extrinsic flexors of the fingers. 22 Perform three maximum repetitions on each side, starting with the dominant upper extremity. The average time to perform each attempt was determined as 5 seconds. During the test, the evaluator will encourage the generation and maintenance of power with a "stronger" verbal command. Finally, the average of the three measurements will be calculated and recorded.
Grip strength | 6 weeks
  It will be evaluated with the JAMAR™ isometric dynamometer (National Institute for Health Research, Southampton), a device recommended by the American Association of Hand Therapists (ASTH). The participant is seated in a chair without an armrest, feet flat on the floor, the shoulder is adducted with neutral rotation, the elbow is positioned at 90° flexion and the forearm is neutral. The JAMAR™ handle is worn in the second position, which allows for balanced activation of the intrinsic and extrinsic flexors of the fingers. 22 Perform three maximum repetitions on each side, starting with the dominant upper extremity. The average time to perform each attempt was determined as 5 seconds. During the test, the evaluator will encourage the generation and maintenance of power with a "stronger" verbal command. Finally, the average of the three measurements will be calculated and recorded.
Grip strength | 12 weeks
  It will be evaluated with the JAMAR™ isometric dynamometer (National Institute for Health Research, Southampton), a device recommended by the American Association of Hand Therapists (ASTH). The participant is seated in a chair without an armrest, feet flat on the floor, the shoulder is adducted with neutral rotation, the elbow is positioned at 90° flexion and the forearm is neutral. The JAMAR™ handle is worn in the second position, which allows for balanced activation of the intrinsic and extrinsic flexors of the fingers. 22 Perform three maximum repetitions on each side, starting with the dominant upper extremity. The average time to perform each attempt was determined as 5 seconds. During the test, the evaluator will encourage the generation and maintenance of power with a "stronger" verbal command. Finally, the average of the three measurements will be calculated and recorded.
Pinch Strength | Baseline
  The individual sits upright on the chair, adducts his shoulder close to his body, and flexes his elbow. For hand and finger grip strengths, one minute intervals are given between each measurement, three measurements are made and the averages are recorded. Measurements; When the individual is in a sitting position, the shoulder is in adduction and neutral rotation, the elbow is in 90 degrees flexion, the forearm is in neutral rotation and supported, and the wrist is in neutral, and it will be repeated 3 times with 30-second breaks. The average of 3 measurements will be taken as the result measurement. The key pinch method will be used in finger pinch strength measurement, and following this measurement, the patient's elbow will be brought to full extension and grip strength will be measured.
Pinch Strength | 6 weeks
  The individual sits upright on the chair, adducts his shoulder close to his body, and flexes his elbow. For hand and finger grip strengths, one minute intervals are given between each measurement, three measurements are made and the averages are recorded. Measurements; When the individual is in a sitting position, the shoulder is in adduction and neutral rotation, the elbow is in 90 degrees flexion, the forearm is in neutral rotation and supported, and the wrist is in neutral, and it will be repeated 3 times with 30-second breaks. The average of 3 measurements will be taken as the result measurement. The key pinch method will be used in finger pinch strength measurement, and following this measurement, the patient's elbow will be brought to full extension and grip strength will be measured.
Pinch Strength | 12 weeks
  The individual sits upright on the chair, adducts his shoulder close to his body, and flexes his elbow. For hand and finger grip strengths, one minute intervals are given between each measurement, three measurements are made and the averages are recorded. Measurements; When the individual is in a sitting position, the shoulder is in adduction and neutral rotation, the elbow is in 90 degrees flexion, the forearm is in neutral rotation and supported, and the wrist is in neutral, and it will be repeated 3 times with 30-second breaks. The average of 3 measurements will be taken as the result measurement. The key pinch method will be used in finger pinch strength measurement, and following this measurement, the patient's elbow will be brought to full extension and grip strength will be measured.
Daily Living Activities | Baseline
  The modified Barthel Activities of Daily Living scale is a questionnaire that measures nutrition, transfer, self-care, sitting on the toilet, washing, walking on a smooth surface, going up and down stairs, dressing, bowel care, and bladder care. The activities are scored according to the degree of ability of the person and the total score determines the degree of addiction.
Daily Living Activities | 6 week
  The modified Barthel Activities of Daily Living scale is a questionnaire that measures nutrition, transfer, self-care, sitting on the toilet, washing, walking on a smooth surface, going up and down stairs, dressing, bowel care, and bladder care. The activities are scored according to the degree of ability of the person and the total score determines the degree of addiction.
Daily Living Activities | 12 week
  The modified Barthel Activities of Daily Living scale is a questionnaire that measures nutrition, transfer, self-care, sitting on the toilet, washing, walking on a smooth surface, going up and down stairs, dressing, bowel care, and bladder care. The activities are scored according to the degree of ability of the person and the total score determines the degree of addiction.
Function | Baseline
  Timed up and go test: Participants will perform certain sequences of movements: getting up from a chair (41 cm height with back support), walking three meters, turning, walking back to the chair, and sitting again. The test will be performed three times and the shortest time (in seconds) will be used for analysis.
Function | 6 week
  Timed up and go test: Participants will perform certain sequences of movements: getting up from a chair (41 cm height with back support), walking three meters, turning, walking back to the chair, and sitting again. The test will be performed three times and the shortest time (in seconds) will be used for analysis.
Function | 12 week
  Timed up and go test: Participants will perform certain sequences of movements: getting up from a chair (41 cm height with back support), walking three meters, turning, walking back to the chair, and sitting again. The test will be performed three times and the shortest time (in seconds) will be used for analysis.
Function (upper extremity) | Baseline
  It consists of 11 items from a 30-item DASH questionnaire designed to assess symptoms and physical and social functions related to upper extremity complaints. Each item is scored on a 1 to 5 scale; A final score between 0 and 100 where 1 indicates "no difficulty" and 5 indicates "extreme difficulty", and a maximum score indicates greater upper extremity dysfunction.
Function (upper extremity) | 6 weeks
  It consists of 11 items from a 30-item DASH questionnaire designed to assess symptoms and physical and social functions related to upper extremity complaints. Each item is scored on a 1 to 5 scale; A final score between 0 and 100 where 1 indicates "no difficulty" and 5 indicates "extreme difficulty", and a maximum score indicates greater upper extremity dysfunction.
Function (upper extremity) | 12 weeks
  It consists of 11 items from a 30-item DASH questionnaire designed to assess symptoms and physical and social functions related to upper extremity complaints. Each item is scored on a 1 to 5 scale; A final score between 0 and 100 where 1 indicates "no difficulty" and 5 indicates "extreme difficulty", and a maximum score indicates greater upper extremity dysfunction.

SECONDARY OUTCOMES:
Balance | Baseline
  Berg Balance Scale: The scale includes 14 increasingly difficult tasks, including changing body position, maintaining a sitting position, maintaining a standing position with and without visual control, standing in a tandem position, standing on one leg, pivoting, reaching forward, lifting objects.
Balance | 6 weeks
  Berg Balance Scale: The scale includes 14 increasingly difficult tasks, including changing body position, maintaining a sitting position, maintaining a standing position with and without visual control, standing in a tandem position, standing on one leg, pivoting, reaching forward, lifting objects.
Balance | 12 weeks
  Berg Balance Scale: The scale includes 14 increasingly difficult tasks, including changing body position, maintaining a sitting position, maintaining a standing position with and without visual control, standing in a tandem position, standing on one leg, pivoting, reaching forward, lifting objects.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, PhD, Principal Investigator — Medipol University
Locations (1):
- Gizem Ergezen, Istanbul, Beykoz, Turkey (Türkiye)